CLINICAL TRIAL: NCT04924673
Title: Study of the Changes in Glycemic Control and Psychological Distress in Diabetic Patients After the Confinement Period Related to the COVID-19 Epidemic
Brief Title: Impact of the COVID-19 Epidemic on Glycemic Balance and the Level of Stress in Diabetic Patients
Acronym: COVIGLYSTRESS
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Collaborators: Pr Pierre-Henri Ducluzeau, University of Tours, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: 35RC20_9780_COVIGLYSTRESS
Record Dates: First submitted 2021-06-10; First posted 2021-06-14 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Diabetes
Keywords: COVID 19; Diabetes; Stress; HbA1c
MeSH Terms: conditions — Diabetes Mellitus; COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective, non-interventional, multicentric study

DETAILED DESCRIPTION:
The rapid spread of the COVID-19 pandemic and the isolation at home implemented in France, creates unprecedented challenges for diabetic patients.

Patients with diabetes have been considered to be at higher risk of infection by the virus, with a greater risk of mortality; this has been a great source of anxiety for them.

It is well known that stress has an impact on plasma glucose levels. The French situation where a general confinement has been decreed over the whole territory (which is not the case for all countries) and for a period of two months, makes it possible to study the impact of this unique situation on stress, sedentary lifestyle, changes in diet and decrease in physical activity. There are no similar experiences described in the literature.

The investigators hypothesize there will be an increase of HbA1c in the coming months.

The main objective is to assess changes in glycemic control in diabetic patients after the confinement period.

The secondary objectives are to:

* Evaluate the prevalence of a state of psychological distress (which could be described as post-traumatic) following this epidemic situation in a population of patients with diabetes and to determine the main characteristics of patients with such a state of psychological distress.
* Study the evolution of the psychological state at a distance from confinement (6 months later) with the same questionnaire.
* Analyze characteristics of lifestyle during confinement: food (snacking), frequency of leaving home, sleep disorders and assess a possible association with variations in HbA1c.

This is an observational, prospective, multicenter study. Participation in the study will be offered to all consecutive patients seen in Diabetes consultations, who meet the selection criteria.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years old)
* Diabetic patient (type 1 or type 2) regardless of their diabetes treatment who experienced complete confinement in their own home, in France.
* Patients who had a measured HbA1 or an estimated HbA1c with a glucose sensor Freestyle libre with a known result, between November 1, 2019 and February 29, 2020.
* Patients agreeing to have their HbA1c measured between May 15 and July 31, 2020.
* Having been informed of the study and not objecting to participating in it

Exclusion Criteria:

- Adults over the age of legal protection (safeguard of justice, curatorship, guardianship), persons deprived of their liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participation in the study will be offered to consecutive diabetic patients (both type 1 and type 2) in Diabetes consultations, who meet the selection criteria; recruitment will be from 11 academic hospitals in France.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-04-22 (Actual)

PRIMARY OUTCOMES:
HbA1c | Baseline
  The change in HbA1c over the first confinement period as compared to the value in early 2020.

SECONDARY OUTCOMES:
Stress | Baseline
  The level of stress as assessed by the GHQ questionnaire and the prevalence of a state of psychological distress (defined by a Likert index in the GHQ test 12 ≥14) both evaluated after the first confinement period in France and then 6 months later, in this population of diabetic patients.

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice BONNET, Principal Investigator — Rennes University Hospital
Locations (11):
- France (11):
  - Rennes University Hospital, Rennes, Brittany Region
  - Centre Hospitalier de l'Agglomération Montargoise, Montargis, Centre-Val de Loire
  - Brest University Hospital, Brest
  - CHU de Dijon, Dijon
  - CHU Grenoble, Grenoble
  - Hospices Civils Lyon, Lyon
  - GHRMSA, Mulhouse
  - CHU Rouen Hôpital Boisguillaume, Rouen
  - CH de Saint Malo, St-Malo
  - CHRU de Tours, Tours
  - Bretagne Atlantique Hospital, Vannes